CLINICAL TRIAL: NCT01404182
Title: Tolerability and Immunogenicity Study of Fluval AB Influenza Vaccine (Trivalent, Seasonal, Active Ingredient Content: 15 μg HA/Strain/0.5 mL) in Adults and Elderly Persons
Brief Title: Tolerability and Immunogenicity Study of Fluval AB Influenza Vaccine in Adults and Elderly Persons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FluvalAB-H-YL2011; 2011-002158-30 (EudraCT Number)
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: seasonal; prevention; influenza; infection; influenza vaccine; vaccine; influenza in humans
MeSH Terms: conditions — Influenza, Human; Infections | interventions — Vaccination; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Influenza vaccination (Experimental): Vaccination with a single dose of Fluval AB influenza vaccine (trivalent, seasonal, active ingredient content: 15 μg HA/0.5mL of seasonal H1N1, H3N2 and B influenza antigens each) and aluminium phosphate gel adjuvant.
  Interventions: Biological: Vaccination with Fluval AB influenza vaccine

INTERVENTIONS:
Biological: Vaccination with Fluval AB influenza vaccine — Vaccination with a single dose of Fluval AB influenza vaccine (trivalent, seasonal, active ingredient content: 15 μg HA/0.5mL of seasonal H1N1, H3N2 and B influenza antigens each) and aluminium phosphate gel adjuvant.
  Other Names: Influenza; Seasonal vaccine; Vaccination; Prevention; Influenza vaccine; Influenza in humans

SUMMARY:
The purpose of this study is to determine the immunogenicity and tolerability of Fluval AB trivalent influenza vaccine in adults and elderly people.

DETAILED DESCRIPTION:
Immunogenicity Objective:

To assess immunogenicity of a single intramuscular (IM) injection of Fluval AB influenza vaccine (trivalent, seasonal, active ingredient content: 15 μg HA/0.5mL of seasonal H1N1, H3N2 and B influenza antigens each), as measured by haemagglutination inhibition (HI) test.

Safety and Tolerability Objectives:

To evaluate safety and tolerability (incidence of adverse events) of a single intramuscular (IM) injection of Fluval AB influenza vaccine (trivalent, seasonal, active ingredient content: 15 μg HA/0.5mL).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years, elderly persons aged over 60 years, both sexes, mentally competent
* Are in good health (as determined by vital signs and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study
* Female volunteers aged 18-60 years (i.e. participants of childbearing potential) with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and not become pregnant for the duration of the study.
* Capability of participants to understand and comply with planned study procedures
* Participants aged above 18 years provide written informed consent prior to initiation of study procedures
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy, breast feeding or positive urine pregnancy test at baseline prior to vaccination. Female subjects who are able to bear children but not willing to use an acceptable contraception method for the duration of the study.
* Known hypersensitivity to eggs, chicken protein, thiomersal, formaldehyde, gentamycin, ciprofloxacin, neomycin or any other component of the vaccine
* History of Guillain-Barré syndrome
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
* Serious disease, such as cancer, autoimmune disease, advanced arteriosclerotic disease, complicated diabetes mellitus, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure
* Immunosuppressive therapy within the past 36 months
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids
* Receipt of immunostimulants,
* Receipt of parenteral immunoglobulin, blood products and/or plasma derivate within the past 3 months
* Suspected or HIV, HBV or HCV infection
* Acute disease and/or axillary temperature ≥37oC within the past 3 days
* Vaccine therapy within the past 4 weeks
* Influenza vaccination (any kind) within the past 6 months
* Experimental drug therapy within the past 4 weeks
* Concomitant participation in another clinical study
* Any condition which, in the opinion of the investigator, may interfere with the evaluation of the study
* Past or current psychiatric disease of the volunteer that upon judgement of the investigator may have effect on the objective decision-making of the volunteer
* Alcohol or drug abuse of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Post vaccination HI antibody titer | 21-28 days following vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions | 21-28 days following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ferenc Tamás, MD, Principal Investigator — Family Doctor's Office Pilisvorosvar; László Sinka, MD, Principal Investigator — Fourmed Gyogyhaz Kft.
Locations (2):
- Hungary (2):
  - Family Doctor's Office, Pilisvörösvár, Pest County
  - Fourmed Gyogyhaz Kft., Veszprém, Veszprém megye